CLINICAL TRIAL: NCT06307769
Title: Examining the Use of the 10-meter Walking Test With Obstacle in Geriatric Individuals.
Brief Title: Ten-meter Walking Test With Obstacle in Geriatric Individuals.
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Birol Onal, Assistant professor, Ataturk University
Other Study IDs: 2024.02.42
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-03

CONDITIONS: Geriatric; Balance
Keywords: Geriatric Individuals, Balance, Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Geriatric Group: balance assessment
- Control Group: balance assessment

SUMMARY:
Balance and fall problems are one of the most common geriatric syndromes in the elderly. Falls are one of the leading factors causing mortality in the elderly. One-third of individuals aged sixty-five and over fall once or more every year. When the causes of death in elderly individuals are examined; Accidents come in fifth place, and 2/3 of these accidents occur due to falls. The frequency of falls increases with age in 22% of individuals between the ages of 65-69. This rate is stated as 31% between the ages of seventy-five and seventy-nine, and 40% between the ages of 80-84.

Geriatric individuals may be at risk of falling in different situations, often inside and outside the home. Falls generally occur more frequently in indoor areas such as bathrooms, kitchens and bedrooms. In these areas, falls caused by potentially dangerous factors such as slippery floors, carpet edges, and high thresholds are more common. A frequent fall occurs when jumping over an obstacle. Factors such as poor balance, vision problems or reduced muscle strength when overcoming obstacles can increase the risk of falling in this situation. The ability of geriatric individuals to overcome obstacles during daily activities is an important factor determining quality of life. Climbing stairs or crossing high thresholds is an important part of daily living activities and poses a risk of falling. Therefore, determining the stair height threshold and assessing obstacle crossing skills should be considered effective measures. When the literature is examined, clinicians generally prefer simpler functional tests because assessments involving disabilities take a long time to be administered, involve some equipment, and also require training to perform the assessment. In the literature, there is currently a version of the functional tests that is applied only by adding obstacles to the timed get up and go test. Thanks to this test, the ability of geriatric individuals to overcome obstacles can be evaluated and people can be trained with this test. For this reason, we wanted to determine the suitability of the 10-meter walking test, which is frequently used in geriatric individuals, when applied with the addition of an obstacle.

DETAILED DESCRIPTION:
Balance and fall frequency in geriatric individuals is an important health problem that occurs as a natural consequence of aging. Factors such as decrease in muscle mass, decrease in bone density and changes in sensory organs with aging can negatively affect balance. This may increase the risk of falls in the geriatric population. Falls can cause serious injuries and loss of independent living skills. Therefore, it is important to evaluate balance and fall risk in geriatric individuals, develop preventive strategies and implement appropriate rehabilitation programs.

Geriatric individuals may be at risk of falling in different situations, often inside and outside the home. Falls generally occur more frequently in indoor areas such as bathrooms, kitchens and bedrooms. In these areas, falls caused by potentially dangerous factors such as slippery floors, carpet edges, and thresholds are more common. Another situation occurs when passing over an obstacle. Factors such as poor balance, vision problems or decreased muscle strength when overcoming obstacles can increase the risk of falling in this situation. The ability of geriatric individuals to overcome obstacles during daily activities is an important factor determining quality of life. Climbing stairs or crossing high thresholds is an important part of daily living activities and poses a risk of falling. Therefore, determining the stair height threshold and assessing obstacle crossing skills should be considered effective measures. When the literature is examined, clinicians generally prefer simpler functional tests because assessments involving disabilities take a long time to be administered, involve some equipment, and also require training to perform the assessment. In the literature, there is currently a version of the functional tests that is applied only by adding obstacles to the timed get up and go test. For this reason, we wanted to determine the suitability of the 10-meter walking test, which is frequently used in geriatric individuals, when applied with the addition of an obstacle.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over,
* For the young adult group, individuals between the ages of 30-65
* Individuals who volunteer to participate in the research,
* Individuals without any neurological disease,
* Individuals who do not have cooperation and communication problems

Exclusion Criteria:

* Those with neurological problems (patients diagnosed with Alzheimer's, Parkinson's, Dementia, MS)
* Those with perceptual problems
* Individuals with cooperation and communication problems will not be included.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consist of 2 groups. The first group is geriatric individuals over the age of 65, and the second group is young healthy adults between the ages of 30-65.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Ten Meter Walk Test | two day
  It is a test used to evaluate walking speed. Participants are instructed to walk at a normal walking pace before starting the test (if they use a device for walking support, they are allowed to walk with it). The clock starts when the participant's foot crosses the line at the beginning of the 10-meter course and stops when it crosses the line at the end of the course. Two measurements are made and the average walking speed is calculated in meters per second (m/s) (1). During the test, the test will also be performed with disabilities by adding 5 and 17 cm obstacles in addition to the original test. In this way, the use of the test applied by adding 5 and 17 cm obstacles will be evaluated in geriatric individuals.

SECONDARY OUTCOMES:
Berg Balance Scale | two day
  BBS was used to evaluate the patients' balance. BBS is a scale consisting of 14 items that evaluates tasks frequently used in daily living activities. Standing from sitting, sitting without support, standing without support, sitting while standing, transfers, standing with eyes closed, standing with legs together, reaching forward while standing, picking up objects from the floor, looking back from both sides, turning 360 degrees, stepping on the step alternately It includes functions such as taking, standing with one foot forward and standing on one leg. Each item is scored between 0-4; 0 indicates that the individual was unable to perform the task, and 4 indicates that the individual was successful in the task.
Functional Reach Test | two day
  During this test, which evaluates the ability to reach forward maximum in a standing position, the participant is asked to reach the furthest distance he can, keeping his arm in 90° flexion, keeping his heels in contact with the ground, without disturbing the parallelism of the arm to the wall, and maintaining his balance. The distance between the shoulder and the fingertip is recorded in cm.
Timed up and go test | two day
  Timed up and go test is used to evaluate mobility and fall risk in elderly people. The test is performed with a comfortable shoe that the patient wears daily, and the patient is allowed to use a walking aid if necessary. The test is performed by recording the time in seconds (sec.) between giving the "go" command while the individual is sitting in the chair, getting up without holding on to the arms of the chair, returning after walking in a predetermined 3-meter area, and sitting on the chair again without support.

CONTACTS AND LOCATIONS:
Overall Officials: Birol Önal, Dr, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Onal B, Kocaman AA. The validity and reliability of the 10-meter walk test with obstacles in community-dwelling older adults. Int J Rehabil Res. 2025 Jun 1;48(2):120-125. doi: 10.1097/MRR.0000000000000665. Epub 2025 Apr 28. PMID 40177963